CLINICAL TRIAL: NCT06184672
Title: Effects of Dry Needling on Latent Myofascial Trigger Points on Vertical Jump Performance in Female Athletes."
Brief Title: Effects of Dry Needling on Vertical Jump Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 008
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: single-blind randomized clinical trial. two groups: intervention group and control group.
Who Masked: Outcomes Assessor
Masking Description: assesor in another isolated room with no possibility of seeing which subjects have been treated or not. Subjects will be informed that they cannot disclose whether they have been needled or not."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): the principal investigator will apply the dry needling technique to those allocated to the experimental group on the latent trigger points diagnosed on the selection phase. They will receive just one session following Hongs protocol.
  Interventions: Other: dry needling
- control group (No Intervention): Subjects in the control group will be asked to wait on the intervention couch for a similar time the ones who received the treatment.

INTERVENTIONS:
Other: dry needling — the area is disinfected by the use of 0.5% chlorhexidine digluconate alcohol solution. The physiotherapist in charge of the intervention uses sterile nitrile gloves, using dry needling needles with dimensions of 0.30 x 50 mm is used. This technique, designed by Hong, applies speed both at the entrance, in order to provoke the local spasm response and at the exit. The inputs and outputs are performed until the REL disappears or until the tolerance threshold of the patient is reached.
  Immediately after performing the puncture, ischemic compression is performed on the treated muscle, in order to decrease the duration and intensity of post-puncture pain. For this, a digital pressure is made to the point where the patient's sensation ceases to be pressure and becomes pain. Once the patient is noted that pain is repeated again the art up to a total of 2 minutes
  Arms: intervention group

SUMMARY:
ChatGPT ChatGPT Injury prevention and performance enhancement have become two of the main goals in every sport. Myofascial Pain Syndrome is primarily caused by myofascial trigger points, which may result in referred pain, stiffness, shortening, and/or muscle weakness.

The aim of this study is to assess the effects of dry needling on latent myofascial trigger points (LTMTP) and its impact on vertical jump height in female volleyball players.

The study is a single-blind, randomized controlled clinical trial conducted on healthy female volleyball practitioners with no lower limb injuries in the last 6 months. Participants must exhibit LMTP in the triceps surae muscles and be familiar with the counter-movement jump (CMJ) test. Subjects will be randomly assigned to either a control group or an intervention group.

DETAILED DESCRIPTION:
This study will be a single-blind, randomized clinical trial conducted in the Department of Invasive Physiotherapy at a private Physiotherapy Clinic in Toledo.

The inclusion criteria are as follows: healthy female volleyball practitioners with no lower limb injuries in the last 6 months, the presence of latent MTPs in the gastrocnemius, and familiarity with performing CMJ tests. Subjects will not be eligible for the study if they have needle phobia, active MTPs in the lower limb, any pathology preventing the use of dry needling, or any pathology preventing the performance of the CMJ test.

Subjects will be randomly assigned to two groups: the intervention group and the control group. Sealed cards containing numbers 1 to 24 in opaque envelopes will be provided, and participants will randomly select a card. Odd-numbered subjects will become part of the control group, while subjects with even numbers will be part of the intervention group.

All subjects must sign a copy of the consent form, which describes and explains the objectives and procedures of the study.

Both groups will undergo a standard warm-up session, including continuous running, dynamic lower limb stretching, and vertical jumps, lasting for 10 minutes (T0). Following the warm-up, the principal investigator will administer the dry needling technique to those assigned to the experimental group. The second measurement will be conducted immediately after the needling technique (T1). Participants in the control group will be instructed to wait on the intervention couch for a comparable duration to those receiving treatment.

The third and fourth assessments will take place in the same clinical setting approximately 72 hours (T3) and 7 days (T4) later, respectively. At each study point, participants will perform 3 CMJ tests. The CMJ-style jumps will be recorded using the high-speed camera of the iPhone 15 (Apple Inc., USA). The My Jump app, validated with a force platform, will calculate the flight time by identifying the subject's takeoff and landing, utilizing an equation from the literature. The best of the three jumps will be recorded. The assessor will be blinded to the allocation group of the participants

ELIGIBILITY:
Inclusion Criteria:

* No lower limb injuries in the last 6 months
* Presence of latent MTPs in gastrocnemius
* Be familiar with performing CMJ tests

Exclusion Criteria:

* Needle phobia
* Presence of active MTPs in the lower limb
* Any pathology that prevented the use of dry needling
* Any pathology that prevented the performance of CMJ test.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-02-08 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
counter movement jump | 4 days
  The subject is in an upright position with the hands at the waist, having to make a vertical jump after a quick countermovement down.
  During knee and hip flexion action, the trunk should remain as straight as possible to avoid any possible influence of trunk extension on lower limb performance.

REFERENCES:
- [Derived] Ladrinan-Maestro A, Sanchez-Infante J, Martin-Vera D, Del-Blanco-Muniz JA, Dominguez-Balmaseda D, Guzman-Pavon MJ, Sanchez-Sierra A. Effects of dry needling on vertical jump performance in female volleyball players. A randomized controlled trial. Front Sports Act Living. 2024 Sep 4;6:1470057. doi: 10.3389/fspor.2024.1470057. eCollection 2024. PMID 39296855